CLINICAL TRIAL: NCT04595396
Title: Gastric Bypass as Metabolic Surgery in Obesity Class 1: a Prospective Study of the Short, Mid and Long Term Results Among Mexicans
Brief Title: Laparoscopic Gastric Bypass as Metabolic Surgery in Obesity Class 1
Status: Completed | Type: Observational
Sponsor: CARLOS ZERRWECK LOPEZ (Other Government)
Responsible Party: Sponsor-Investigator, CARLOS ZERRWECK LOPEZ, Professor and Head of Department., Hospital General Tlahuac
Organization: Hospital General Tlahuac (Other Government)
Other Study IDs: CONBIOETICA09-CEI-001-20160404
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Type2 Diabetes; Bariatric Surgery Candidate; Laparoscopic Gastric Bypass; Obesity
Keywords: bariatric surgery; obesity class 1; metabolic surgery; laparoscopic gastric bypass; type-2 diabetes mellitus
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic Gastric Bypass — The LGBP was performed using a classic Roux-en-Y procedure. Briefly, a gastric pouch of 30-50 cc was constructed with an antecolic calibrated gastro-jejunal anastomosis (mechanical anastomosis using a 2.5 mm load). The biliary and alimentary limbs measured ≈70 cm and ≈150 cm, respectively, and the jejuno-jejunal anastomosis was also performed in a latero-lateral fashion (mechanical anastomosis using a 2.5 mm load). Mesenteric defects were closed with running non-absorbable sutures and the omentum was divided in every case
  Other Names: Roux-en-y gastric bypass

SUMMARY:
Prospective study including Mexican patients diagnosed with type 2 diabetes and class 1 obesity, undergoing laparoscopic gastric bypass. The objective was to determine short, mid-and long-term outcomes (weight loss, metabolic, morbidity and diabetes remission). A subanalysis was included, based on preoperative usage of one (Group A) or more antidiabetics ± insulin (Group B).

ELIGIBILITY:
Inclusion criteria Any sex >18 years-old <60 years-old Class 1 obesity (BMI 30-34.9 kg/m2) Type-2 diabetes mellitus diagnosis (with or without medication) Submitted to laparoscopic gastric bypass

Exclusion criteria Other bariatric surgery Revisional surgery Incomplete charts

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mexican patients with T2DM submitted to laparoscopic gastric bypass
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 months
  Measure: weight (kilograms)
Weight Loss | 24 months
  Measure: weight (kilograms)
Weight Loss | 36 months
  Measure: weight (kilograms)
Weight Loss | 12 months
  Measure: Body Mass Index
Weight Loss | 24 months
  Measure: Body Mass Index
Weight Loss | 36 months
  Measure: Body Mass Index
Weight Loss | 12 months
  Measure: % excess weight loss
Weight Loss | 24 months
  Measure: % excess weight loss
Weight Loss | 36 months
  Measure: % excess weight loss
Weight Loss | 12 months
  Measure: % total weight loss
Weight Loss | 24 months
  Measure: % total weight loss
Weight Loss | 36 months
  Measure: % total weight loss

SECONDARY OUTCOMES:
Complete Diabetes Remission | 12 months
  Definition: no antidiabetic drugs while on glucose <100 mg/dl and HbA1C% <6
Complete Diabetes Remission | 24 months
  Definition: no antidiabetic drugs while on glucose <100 mg/dl and HbA1C% <6
Complete Diabetes Remission | 36 months
  Definition: no antidiabetic drugs while on glucose <100 mg/dl and HbA1C% <6
Late complications | After 30 days from surgery
  Complications requiring re-admssion / re-operation
Early complications | First 30 days after surgery
  Complications requiring re-admssion / re-operation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Tlahuac, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cevallos L, Rodriguez FM, Herrera A, Sepulveda EM, Donatini G, Guilbert L, Zerrweck C. Metabolic Surgery and Class 1 Obesity (< 35 kg/m2): a Prospective Study with Short-, Mid-, and Long-term Results Among Latinos. Obes Surg. 2021 Jun;31(6):2401-2409. doi: 10.1007/s11695-021-05275-3. Epub 2021 Feb 17. PMID 33598844